CLINICAL TRIAL: NCT01552421
Title: The Effect of Transvaginal vs. Conventional Laparoscopic Cholecystectomy on the Postoperative Course
Acronym: TRAVAKOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For logistic reasons in the department and due to very low inclusion rates.
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other); University Hospital, Gentofte, Copenhagen (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anders Meller Donatsky, MD, PhD-student, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOTES02
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Cholecystolithiasis; Surgery; Pain
Keywords: Cholecystectomy; Natural Orifice Transluminal Endoscopic Surgery; Transvaginal cholecystectomy; Postoperative outcome
MeSH Terms: conditions — Cholecystolithiasis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TV NOTES cholecystectomy (Active Comparator): Participants randomized to TV NOTES cholecystectomy
  Interventions: Procedure: TV NOTES cholecystectomy
- Laparoscopic cholecystectomy (No Intervention): Participants randomized to laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: TV NOTES cholecystectomy — Transvaginal NOTES cholecystectomy
  Arms: TV NOTES cholecystectomy

SUMMARY:
Uncomplicated laparoscopic cholecystectomy will in most patients result in moderate to severe pain until the first postoperative day. This will subside during the second and third postoperative day [1]. A feeling of low general well-being will also be present until the first postoperative day and subside during the next couple of days [2].

To achieve faster recovery after laparoscopic interventions it has been shown that a reduction in the size of laparoscopic ports and thereby incisions can reduce postoperative pain [3,4].

A new minimal invasive surgical technique is based on the principle of completely eliminating the use of ports through the abdominal wall. This new technique is called Natural Orifice Transluminal Endoscopic Surgery (NOTES) and is defined by acquiring minimal invasive access to the abdominal cavity through the body's natural openings like the mouth and stomach, anus, urethra and vagina. With the NOTES technique one can completely avoid incisions in the abdominal wall and thereby reduce the surgical trauma. The benefits of this technique is a reduction of postoperative pain, elimination of incisional hernias, prevention of wound infections, reduction of peritoneal adherence formation, achieving a faster recovery and a better cosmetic result [7,8].

The most documented and well-described way for gaining NOTES access to the abdominal cavity is through the vagina, transvaginal (TV). TV NOTES has mainly been used for cholecystectomy because of the direct line of vision to the upper abdomen and gallbladder that is achieved through this opening.

Compilation of results show that TV NOTES cholecystectomy can be implemented with low complication rates [20-22]. One retrospective case-control and one prospective observational study report less postoperative pain, reduced consumption of analgesics and faster recovery for TV NOTES compared to conventional laparoscopic cholecystectomy [23,24]. To date there are no systematic prospective randomized data on whether or not TV NOTES cholecystectomy leads to a better surgical outcome.

In the present study the postoperative course after TV NOTES cholecystectomy will be compared to laparoscopic cholecystectomy in a prospective randomized and blinded trial. The outcome of the randomization between the two surgical techniques will be blinded to patient and the nurse staff for the first 72 hours after the operation. The primary outcome parameter will be postoperative pain score during the first 24 hours. Secondary outcome parameters are postoperative pain score for the first 72 hours, fatigue, well-being, nausea, consumption of analgesics, complications, cosmetic result and sexual function.

The hypothesis being that TV NOTES cholecystectomy gives less postoperative pain, fatigue and nausea, a reduction in analgesics and a better cosmetic result and general well-being than conventional 4 port laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
BACKGROUND:

Uncomplicated laparoscopic cholecystectomy will in most patients result in moderate to severe pain up until the first postoperative day. This will subside during the second and third postoperative day [1]. A feeling of low general well-being will also be present up until the first postoperative day and subside during the next couple of days [2].

To achieve faster recovery after laparoscopic interventions it has been shown that a reduction in the size of laparoscopic ports and thereby incisions can reduce postoperative pain [3,4]. Whether a further reduction of postoperative pain can be achieved by limiting the number of laparoscopic ports through the abdominal wall to a single one with Single Incision Laparoscopic Surgery (SILS) remains to be determined [5,6].

A new minimal invasive surgical technique is based on the principle of completely eliminating the use of ports through the abdominal wall. This new technique is called Natural Orifice Transluminal Endoscopic Surgery (NOTES) and is defined by acquiring minimal invasive access to the abdominal cavity through the body's natural openings like the mouth and stomach, anus, urethra and vagina. With the NOTES technique one can completely avoid incisions in the abdominal wall and thereby further reduce the surgical trauma. The benefits of this technique is a reduction of postoperative pain, elimination of incisional hernias, prevention of wound infections, reduction of peritoneal adherence formation, achieving a faster recovery and a better cosmetic result [7,8].

The most documented and well-described way for gaining NOTES access to the abdominal cavity is through the vagina, transvaginal (TV). There are several reasons for this. First of all the technique for gaining TV access to the abdominal cavity is already being used in gynaecology, where culdoscopy was first described in the literature nearly 100 years ago [9]. A diagnostic procedure for infertility that can be used in an outpatient setting [10-12]. Similarly, transvaginal ports have been used in gynaecology as a substitute for abdominal ports [13,14]. Thus there is already a well proven and established technique for obtaining transvaginal access to the abdominal cavity. Secondly it is easy to ensure a secure surgical closure of the point of entry under direct visualization with basic suturing instruments. And lastly the risk of contamination and infection is minimal when performing TV procedures [15].

TV NOTES has mainly been used for cholecystectomy because of the direct line of vision to the upper abdomen including the liver and gallbladder that is achieved through this body opening. For the same reason it is possible to use the same surgical dissection technique and rigid instruments that is used when performing conventional laparoscopic or SILS cholecystectomies.

Questionnaire surveys have shown that there is a general interest for TV NOTES in the public, where between 33-68 % of women surveyed preferred TV NOTES to conventional laparoscopy [16-18].

In a German national database called German NOTES Registry (GNR) more than 900 transvaginal procedures have been registered. Compilation of results from the GNR and other human series and multicenter trials have shown that TV NOTES cholecystectomy can be implemented with low complication rates [19-21]. One retrospective case-control and one prospective observational study report less postoperative pain, reduced consumption of analgesics and faster recovery for TV NOTES cholecystectomy compared to conventional laparoscopic cholecystectomy [22,23]. To date there are no systematic prospective randomized data on whether or not TV NOTES cholecystectomy leads to a better surgical outcome in regards to pain, well-being etc. than conventional laparoscopic cholecystectomy.

STUDY AIM:

The aim of the study is in a prospective randomized blinded design to compare the postoperative course and outcome of TV NOTES and conventional laparoscopic cholecystectomy.

HYPOTHESIS:

TV NOTES cholecystectomy gives less postoperative pain, fatigue and nausea, reduces analgesic consumption and gives a better cosmetic result and well-being than conventional 4 port laparoscopic cholecystectomy.

TRIAL PARTICIPANTS:

Trial participants will be recruited among women between 40-75 years referred to laparoscopic cholecystectomy due to symptomatic gallstones or gallstone induced mild pancreatitis and ultrasonography confirmed gallstones.

METHOD:

Statistics:

The primary outcome measure "cumulated pain score during mobilisation for the first 72 postoperative hours" has been used for power calculation. In a previous study the mean for this parameter measured on the visual analogue scale (VAS) for laparoscopic cholecystectomy have been found to be 143 mm (standard deviation 95,7 mm) [2]. Since the pain sensation after laparoscopic cholecystectomy is somatic in origin a MERIDIF of 60% (86mm) have been chosen. Type I and type II errors have been set to 0,05 and 0,20 respectively. This gives a total number of 42 participants with 21 in allocated to either group. To account for potential dropouts and the lack of Gaussian distribution for VAS data there will be included a total of 60 participants with 30 allocated to either group.

Non-parametric statistics with Fisher´s exact test, Mann-Whitney test and confidence intervals will be used where appropriate. P < 0,05 will be considered statistical significant. Drop-outs will be replaced by new participants until a minimum of 30 participants have been included in either group. Data will be analysed with intention-to treat and per-protocol and the results of both methods will be published.

In the TV NOTES group the use of at least one 5mm trans-abdominal port will be considered as a conversion to conventional laparoscopic surgery and will analysed as such. The use of one Minilap instrument in the TV NOTES group will not be considered as a conversion to laparoscopy and the participant will remain in the TV NOTES group for both the intention-to-treat and the per-protocol analyses. Participants with severe intra-operative complications will be excluded from the analyses but will be described separately in the publication.

Randomization:

Participants will be randomized to either TV NOTES cholecystectomy or conventional laparoscopic 4 port cholecystectomy. The randomization will be performed shortly before the operation commences using the envelope method by the operating surgeon. All procedures will be performed by the same surgeon at University Hospital Gentofte/Herlev, Copenhagen, Denmark.

Blinding:

The trial is patient and observer blinded to the allocation of the randomization for the first 72 hours of the postoperative course. Operating room staff and surgeons will not participate in any way in the follow-up for the first 72 postoperative hours.

Participants in both groups will receive the same surgical dressing on the abdomen after the procedure. Both groups will thus be bandaged as if after a conventional 4 port laparoscopic cholecystectomy with a total of 4 dressing strips. In the TV NOTES group these dressings will be stained red to simulate light seepage from the "wound". These dressings are obligatory for the first 72 postoperative hours.

Informed consent:

The participants will receive oral and written information about the trial, its purpose and potential benefits and risks. Participants will be informed that it is voluntary to participate at that they at any time can withdraw their consent to participate in the trial without it having any implications on present or future treatment. Written consent to participate in the trial will be obtained before enrolment. National guidelines from the Danish National Committee on Biomedical Research Ethics concerning informed content will be followed.

Any information or medical considerations concerning the individual participant obtained as part of the trial will be accessible to the participant.

ETHICAL CONSIDERATIONS:

TV NOTES cholecystectomy are based on well-established surgical techniques such as laparoscopy/SILS and culdotomy. Complication types and rates for TV NOTES cholecystectomy are well described in the literature and are comparable to that of conventional laparoscopic cholecystectomy. Considering the advantages and theoretical benefits this new technique has to offer combined with the preliminary retrospective and non-randomized results we find it ethical to conduct a randomized controlled blinded trial where the benefits of TV NOTES cholecystectomy outweighs the potential risks involved.

LAW AND APPROVAL:

The trial will be carried out according to the Helsinki Declaration II and under the Acts of the Danish Council of Ethics and information concerning the participants will be protected in accordance to the regulations set by the Danish Protection Agency. The trial will be approved by the Danish National Committee on Biomedical Research Ethics, the Danish Protection Agency and ClinicalTrials.gov before it is commenced.

FUNDING:

This trial is part of a PhD-study initiated by the trial investigators. Salaries are funded through grants obtained from the University of Copenhagen, Herlev Hospital Research Council, Capitol Region of Denmark Research Foundation for Health Research and private foundations. Operating costs are founded through grants from private foundations. There are no commercial interests in or financial support for the project.

PUBLICATION:

After the trial have been completed both positive and negative result will be published in an internationally recognised scientific journal. The primary investigator in this trial will be first-author and the co-investigators co-authors according to the Vancouver Group criteria (www.icmje.org).

ELIGIBILITY:
Inclusion Criteria:

* Booked for cholecystectomy due to symptomatic gallstones or gallstone induced mild pancreatitis.
* Woman.
* Between 18 - 70 years old.
* ASA classification I, II or III.
* BMI < 30 kg/m2.
* Written informed consent.

All of the inclusion criteria must be met before inclusion in the study.

Exclusion Criteria:

* Expected poor compliance.
* Previous cholecystitis or moderate to severe pancreatitis.
* Culdotomy contraindicated.
* Previous laparoscopic surgery or open surgery on vagina, uterus, fallopian tubes or ovaries. Except laparoscopic sterilisation.
* Pregnancy or breastfeeding.
* Daily consumption of any analgesic for one month prior to surgery or intermittent use of opioids.
* Ongoing treatment with Monoamine Oxidase Inhibitors or Tricyclic antidepressants.
* Known with any type of inflammatory bowel disease.
* Known with chronic diseases that are known to cause pain sensations.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cumulated postoperative pain with visual analogue scale (VAS) | 72 hours
  Postoperative pain will be measured with VAS, 3 hours after the operation as well as on the first, second and third postoperative day. Pain score will be assessed at rest and during mobilization from supine to erect posture. Based on these assesments a cumulated overall pain score for the first 72 postoperative hours will be calculated by adding the respective scores for each participant.

SECONDARY OUTCOMES:
Postoperative fatigue | 72 hours
  Postoperative fatigue will be measured on a scale from 0 (no fatigue) to 10 (severe fatigue) 3 hours post surgery and on postoperative day 1, 2 and 3.
Postoperative well-being | 72 hours
  Well-being will be measured with VAS 3 hours post surgery and on postoperative day 1, 2 and 3.
Postoperative nausea | 72 hours
  Nausea will be measured with VRS 3 hours post surgery and on postoperative day 1, 2 and 3.
Postoperative vomiting | 72 hours
  Total number of times the participant have been vomiting 3 hours post surgery and on postoperative day 1, 2 and 3.
Postoperative analgesic and antiemetic consumption | 72 hours
  All participants will be given oral Paracetamol 1g four times a day and Ibuprofen 400 mg three times a day for the first 72 postoperative hours. Any need for additional analgesics besides this will be registered. Consumption of antiemetics will be registered.
Postoperative complications | 1 year
  Any postoperative complications will be registered during the participants admission and on follow-up 28 days (+/- 2 days) and 12 months (+/- 14 days) after surgery
Cosmetic result | 1 year
  Participants will be requested to score their satisfaction with the cosmetic result on a scale from 0 (no scarring) to 10 (severe scarring)28 days (+/- 2 days) and 12 months (+/- 14 days) after surgery.
Sexual function and dyspareunia | 1 year
  Participants are requested to fill in the questionnaire Female Sexual Function Index (FSFI) on sexual function and dyspareunia 28 days (+/- 2 days) and 12 months (+/- 14 days) after surgery.
Postoperative hospitalization | Until the individual participant is discharged from the hospital
  The time from admission to discharge from the hospital is recorded.
Surgical details | Intra-operative
  Details about the technical aspects of performing TV NOTES cholecystectomy is recorded during and immediate after surgery.
Early postoperative pain with VAS | 24 hours
  Early overall postoperative pain measured with VAS, 3 hours after the operation as well as on the first postoperative day. Pain score will be assessed at rest and during mobilization from supine to erect posture.
Late postoperative pain measured with VRS | 48 hours
  Late postoperative pain measured with VRS on the second and third postoperative day. Pain score will be assessed at rest and during mobilization from supine to erect posture.
Early pain localization | 24 hours
  Pain localization (abdominal wall, intra-abdominal or shoulder pain) will be measured with VRS, 3 hours postoperatively as well as on the first postoperative day.
Late pain localization | 48 hours
  Pain localization (abdominal wall, intra-abdominal or shoulder pain) will be measured with VRS, on the second and third postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Meller Donatsky, MD, Principal Investigator — Department of Surgical Gastroenterology, Herlev Hospital; Lars Nannestad Jørgensen, MD, DSc, Prof., Study Chair — Department of Surgery K, Bispebjerg Hospital, University of Copenhagen; Sami Assaadzadeh, MD, Study Chair — Department of Surgical Gastroenterology, Herlev Hospital; Jacob Rosenberg, MD, DSc, Prof., Study Chair — Department of Surgical Gastroenterology, Herlev Hospital, University of Copenhagen; Peter Vilmann, MD, DSc, Prof., Study Chair — Department of Surgical Gastroenterology, Herlev Hospital, University of Copenhagen; Søren Meisner, MD, Study Chair — Department of surgery K, Bispebjerg Hospital
Locations (1):
- Departement of Surgical Gastroenterology, Gentofte Hospital, Gentofte Municipality, Denmark